CLINICAL TRIAL: NCT01494545
Title: Performance Evaluation of DAILIES® TOTAL1™ in First Time Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-347-C-016
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Myopia
Keywords: DAILIES TOTAL1; Alcon; contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delefilcon A (Experimental): Delefilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for two weeks. A new pair was inserted each day.
  Interventions: Device: Delefilcon A contact lens

INTERVENTIONS:
Device: Delefilcon A contact lens — Silicone hydrogel contact lens CE-marked for single use, daily disposable wear
  Other Names: DAILIES® TOTAL1™

SUMMARY:
The purpose of this study was to evaluate the performance of DAILIES® TOTAL1™ in first time contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* No previous contact lens experience or attempt to try contact lenses (neophyte).
* Willing to wear study lenses for at least 8 hours a day for at least 5 days a week.
* Use spectacle lenses for vision correction.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* 45 years or older.
* Prior wear experience with rigid or soft contact lenses.
* Systemic or ocular disease or disorder that would negatively affect the conduct or outcome of the study.
* History of ocular surgery/trauma within the last six months.
* Pregnant or nursing women.
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from study centers in Europe.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | Delefilcon A
Started | 102
Completed | 92
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled participants who were dispensed study product.
Arm/Group | Delefilcon A
Number analyzed (Participants) | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 24.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Initial Comfort
Description: Initial comfort was rated by the participant and recorded on a questionnaire at time of lens dispense. Initial comfort was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 1
Population: This reporting group includes all enrolled and dispensed participants, minus major protocol deviations as determined by review.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale | 8.6 (1.3)

2. Primary Outcome: Comfort at Insertion by Visit
Description: Comfort at insertion was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Comfort at insertion was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.6 (1.3)
  Day 14 | 8.8 (1.2)

3. Primary Outcome: Comfort During the Day by Visit
Description: Comfort during the day was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Comfort during the day was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.7 (1.3)
  Day 14 | 8.9 (1.0)

4. Primary Outcome: Comfort at End of Day by Visit
Description: Comfort at end of day was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Comfort at end of day was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 7.5 (1.8)
  Day 14 | 7.9 (1.5)

5. Primary Outcome: Overall Comfort by Visit
Description: Overall comfort was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Overall comfort was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.5 (1.2)
  Day 14 | 8.7 (1.0)

6. Primary Outcome: Initial Quality of Vision
Description: Initial quality of vision was rated by the participant and recorded on a questionnaire at time of lens dispense. Initial quality of vision was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale | 8.7 (1.1)

7. Primary Outcome: Quality of Vision at Insertion by Visit
Description: Quality of vision at insertion was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Quality of vision at insertion was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.7 (1.2)
  Day 14 | 9.0 (1.2)

8. Primary Outcome: Quality of Vision During the Day by Visit
Description: Quality of vision during the day was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Quality of vision during the day was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.9 (1.2)
  Day 14 | 8.9 (1.1)

9. Primary Outcome: Quality of Vision at End of Day by Visit
Description: Quality of vision at end of day was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Quality of vision at end of day was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.3 (1.5)
  Day 14 | 8.3 (1.4)

10. Primary Outcome: Overall Quality of Vision by Visit
Description: Overall quality of vision was rated by the participant and recorded on a questionnaire as a single, retrospective evaluation of the previous week of lens wear. Overall quality of vision was rated on a 10-point scale (1=poor to 10=excellent) as a single assessment for both eyes.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 7 | 8.8 (1.1)
  Day 14 | 8.8 (1.1)

11. Primary Outcome: Average Comfortable Daily Wear Time by Visit
Description: Average comfortable daily wear time was reported by the participant as a single, retrospective evaluation of the previous week of wear.
Time Frame: Day 7, Day 14
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Hours
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Hours
  Day 7 | 10.3 (3.2)
  Day 14 | 10.4 (2.8)

12. Primary Outcome: Likert Statement: These Contact Lenses Were so Comfortable That I Don't Feel Anything.
Description: The participant indicated agreement/disagreement with the statement by using a 4-point scale: 2=Strongly Agree; 1=Agree; -1=Disagree; -2=Strongly Disagree. A single assessment was made for both eyes.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 17.4
  Agree | 43.5
  Disagree | 37.0
  Strongly Disagree | 2.2

13. Primary Outcome: Likert Statement: These Contact Lenses Were so Comfortable That I Barely Felt Anything.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 19.8
  Agree | 68.1
  Disagree | 12.1
  Strongly Disagree | 0.0

14. Primary Outcome: Likert Statement: These Contact Lenses Felt so Comfortable That I Forgot I Was Wearing Them.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 18.5
  Agree | 45.7
  Disagree | 33.7
  Strongly Disagree | 2.2

15. Primary Outcome: Likert Statement: These Contact Lenses Are Perfect for When I Choose Not to Wear my Eye Glasses.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 45.7
  Agree | 47.8
  Disagree | 5.4
  Strongly Disagree | 1.1

16. Primary Outcome: Likert Statement: I Liked These Contact Lenses so Much That I Will Recommend Them to my Friends.
Description: The participant indicated agreement/disagreement with the statement by using a 4-point scale: 22=Strongly Agree; 1=Agree; -1=Disagree; -2=Strongly Disagree. A single assessment was made for both eyes.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 41.3
  Agree | 54.3
  Disagree | 4.3
  Strongly Disagree | 0.0

17. Primary Outcome: Likert Statement: Overall, my Vision is Better With These Contact Lenses Compared to my Eye Glasses.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 22.8
  Agree | 44.6
  Disagree | 30.4
  Strongly Disagree | 2.2

18. Primary Outcome: Likert Statement: At the End of the Day my Vision is Better With These Contacts Lenses Compared to my Eye Glasses.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 9.8
  Agree | 35.9
  Disagree | 50.0
  Strongly Disagree | 4.3

19. Primary Outcome: Likert Statement: My Peripheral Vision is Better With These Contact Lenses Than With my Eye Glasses.
Description: as for outcome 12
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 46.7
  Agree | 45.7
  Disagree | 7.6
  Strongly Disagree | 0.0

20. Secondary Outcome: Lens Surface Characteristics: Dry Areas/Non-wetting
Description: The investigator assessed the surface of the contact lens while the lens was on the participant's eye for dry areas/non-wetting: 0=None; 1=Very Slight; 2-Slight; 3=Moderate; 4=Severe. Assessments were made individually (by eye) and binocularly (both eyes together).
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Groups:
- Delefilcon A, Right Eye: Delefilcon A contact lenses worn in right eye on a daily wear, daily disposable basis for two weeks. A new lens was inserted each day.
- Delefilcon A, Left Eye: Delefilcon A contact lenses worn in left eye on a daily wear, daily disposable basis for two weeks. A new lens was inserted each day.
- Delefilcon A, Both Eyes: Delefilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for two weeks. A new pair was inserted each day.
Arm/Group | Delefilcon A, Right Eye | Delefilcon A, Left Eye | Delefilcon A, Both Eyes
Number analyzed (Participants) | 92 | 92 | 92
Number analyzed (eyes) | 92 | 92 | 184
Percentage of eyes
  None | 85.9 | 81.5 | 83.7
  Very Slight | 13.0 | 15.2 | 14.1
  Slight | 1.1 | 3.3 | 2.2
  Moderate | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0

21. Secondary Outcome: Lens Surface Characteristics: Dry Areas/Non-Wetting
Description: as for outcome 20
Time Frame: Day 7
Population: as for outcome 1
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Delefilcon A, Right Eye | Delefilcon A, Left Eye | Delefilcon A, Both Eyes
Number analyzed (Participants) | 92 | 92 | 92
Number analyzed (eyes) | 92 | 92 | 184
Percentage of eyes
  None | 81.1 | 82.2 | 81.7
  Very Slight | 15.6 | 15.6 | 15.6
  Slight | 3.3 | 2.2 | 2.8
  Moderate | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0

22. Secondary Outcome: Lens Surface Characteristics: Dry Areas/Non-Wetting
Description: as for outcome 20
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Delefilcon A, Right Eye | Delefilcon A, Left Eye | Delefilcon A, Both Eyes
Number analyzed (Participants) | 92 | 92 | 92
Number analyzed (eyes) | 92 | 92 | 184
Percentage of eyes
  None | 77.2 | 76.1 | 76.6
  Very Slight | 19.6 | 23.9 | 21.7
  Slight | 3.3 | 0.0 | 1.6
  Moderate | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Duration of Overall Training Time
Description: The investigator recorded the time it took for the patient to insert both lenses and remove both lenses, not including instructions.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Minutes
  Insertion time | 6.926 (6.558)
  Removal time | 6.806 (7.872)

24. Secondary Outcome: Investigator's Satisfaction With Lens Fit by Visit
Description: The investigator considered the factors that relate to a well-fitted contact lens, including good centration, adequate movement, and complete corneal coverage, and rated his/her satisfaction with the contact lens fit on 10-point scale, with 1 being not at all satisfied and 10 being very satisfied.
Time Frame: Day 1, Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 1 | 9.2 (0.9)
  Day 7 | 9.3 (0.9)
  Day 14 | 9.3 (0.8)

25. Secondary Outcome: Investigator's Overall Impression of Surface Wettability by Visit
Description: The investigator rated his/her overall impression of the surface wettability of the contact lens on a 10-point scale (1=poor to 10=excellent).
Time Frame: Day 1, Day 7, Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Units on a scale
  Day 1 | 9.3 (0.9)
  Day 7 | 9.3 (1.0)
  Day 14 | 9.3 (1.0)

26. Secondary Outcome: Investigator's Rating of Ease of Fit
Description: The investigator indicated agreement/disagreement with the statement, "The study lenses were easy to fit for this subject," by using a 4-point scale: 1=Strongly Agree; 2=Agree; 3=Disagree; 4=Strongly Disagree.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Strongly Agree | 75.0
  Agree | 22.8
  Disagree | 2.2
  Strongly Disagree | 0.0

27. Primary Outcome: Likert Statement: Compared to my Eye Glasses, my Vision With These Contact Lenses is:
Description: The participant indicated overall satisfaction/dissatisfaction with the contact lenses using a 5-point scale: 2=Much Better; 1=A Little Better; 0=Same; -1=A Little Worse; -2=Much Worse. A single assessment was made for both eyes.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Much Better | 21.7
  A Little Better | 41.3
  Same | 22.8
  A Little Worse | 14.1
  Much Worse | 0.0

28. Primary Outcome: Likert Statement: I am Interested in Purchasing These Contact Lenses.
Description: The participant indicated purchase intent using a 4-point scale: 2=Very Interested; 1=Interested; -1=Not Interested; -2=Very Disinterested. A single assessment was made for both eyes.
Time Frame: Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Delefilcon A
Number analyzed (Participants) | 92
Percentage of participants
  Very Interested | 28.3
  Interested | 64.1
  Not Interested | 7.6
  Very Disinterested | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study from informed consent signature until last follow-up visit.
Description: This reporting group includes all enrolled participants who were dispensed study product.
Arm/Group | Delefilcon A
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.